CLINICAL TRIAL: NCT04072302
Title: A Two-part, Randomized, Double-blind, Placebo-controlled, Single-center Study to Evaluate the Safety and Causal Prophylactic Efficacy of KAF156 in a Controlled Human Malaria Challenge Model
Brief Title: Safety and Causal Prophylactic Efficacy of KAF156 in a Controlled Human Malaria Challenge Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CKAF156X2202
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Malaria
Keywords: Malaria; KAF156; P. falciparum
MeSH Terms: conditions — Malaria | interventions — ganaplacide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- KAF156 800 mg pre-challenge (Experimental): Single dose 800 mg KAF156 oral administration in healthy subjects, prior to exposure to P. falciparum sporozoite-infected mosquitos
  Interventions: Drug: KAF156
- Placebo 800 mg pre-challenge (Placebo Comparator): Single dose 800 mg placebo oral administration in healthy subjects, prior to exposure to P. falciiparum sporozoite-infected mosquitos
  Interventions: Drug: Placebo
- KAF156 800 mg post-challenge (Experimental): Single dose 800 mg KAF156 oral administration in heatlhy subjects, after exposure to P. falciparum sporozoite-infected mosquitos
  Interventions: Drug: KAF156
- Placebo 800 mg post-challenge (Placebo Comparator): Single dose 800 mg placebo oral administration in heatlhy subjects, after exposure to P. falciparum sporozoite-infected mosquitos
  Interventions: Drug: Placebo
- KAF156 300 mg post-challenge (Experimental): Single dose 300 mg KAF156 oral administration in heatlhy subjects, after exposure to P. falciparum sporozoite-infected mosquitos
  Interventions: Drug: KAF156
- Placebo 300 mg post-challenge (Placebo Comparator): Single dose 300 mg placebo oral administration in heatlhy subjects, after exposure to P. falciparum sporozoite-infected mosquitos
  Interventions: Drug: Placebo
- KAF156 100 mg post-challenge (Experimental): Single dose 100 mg KAF156 oral administration in heatlhy subjects, after exposure to P. falciparum sporozoite-infected mosquitos
  Interventions: Drug: KAF156
- Placebo 100 mg post-challenge (Placebo Comparator): Single dose 100 mg placebo oral administration in heatlhy subjects, after exposure to P. falciparum sporozoite-infected mosquitos
  Interventions: Drug: Placebo
- KAF156 20 mg post-challenge (Experimental): Single dose 20 mg KAF156 oral administration in heatlhy subjects, after exposure to P. falciparum sporozoite-infected mosquitos
  Interventions: Drug: KAF156
- Placebo 20 mg post-challenge (Placebo Comparator): Single dose 20 mg Placebo oral administration in heatlhy subjects, after exposure to P. falciparum sporozoite-infected mosquitos
  Interventions: Drug: Placebo
- KAF156 50 mg post-challenge (Experimental): Single dose 50 mg KAF156 oral administration in heatlhy subjects, after exposure to P. falciparum sporozoite-infected mosquitos
  Interventions: Drug: KAF156
- Placebo 50 mg post-challenge (Placebo Comparator): Single dose 50 mg Placebo oral administration in heatlhy subjects, after exposure to P. falciparum sporozoite-infected mosquitos
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KAF156 — 100 mg tablet, 20 mg tablet, 50 mg tablet
  Arms: KAF156 100 mg post-challenge; KAF156 20 mg post-challenge; KAF156 300 mg post-challenge; KAF156 50 mg post-challenge; KAF156 800 mg post-challenge; KAF156 800 mg pre-challenge
Drug: Placebo — 100 mg tablet, 20 mg tablet, 50 mg tablet
  Arms: Placebo 100 mg post-challenge; Placebo 20 mg post-challenge; Placebo 300 mg post-challenge; Placebo 50 mg post-challenge; Placebo 800 mg post-challenge; Placebo 800 mg pre-challenge

SUMMARY:
This study is designed to investigate the safety and causal prophylactic efficacy of KAF156 in healthy subjects using a controlled human malaria infection model.

ELIGIBILITY:
Inclusion Criteria:

- Healthy male subjects,aged 18 to 40 years of age included and in good health as determined by past medical history, physical examination, vital signs, ECG, and laboratory tests

Exclusion Criteria:

* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
* Known history or current clinically significant ECG abnormalities or arrhythmias.
* Symptoms, physical signs and laboratory values suggestive of systemic disorders including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric, or other conditions which could interfere with the interpretation of the study results or compromise the health of the subjects.
* Sexually active males must use a condom during intercourse while taking drug and for al least 4 weeks after stopping study medication and should not father a child during this period.
* History of malaria or residence in a malaria-endemic area over a period of 6 months before study entry. - Any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk or render the subject unable to meet requirements of the protocol.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Number of subjects with parasitemia after single dose oral administration of KAF156 either prior to, or following, exposure to P. falciparum sporozoite-infected mosquitoes | From Day 1 to Day 43
  The number of subjects that became infected with malaria at each dose
Relationship between pharmacokinetics (i.e., Maximum Plasma Concentration [Cmax], Area Under Curve [AUC]) of KAF156 and number of subjects with parasitemia, after oral administration of single descending doses of KAF156 in healthy subjects with CHMI | From Day 1 to Day 43
  The exposure-response relationship of KAF156 was explored in a PK/PD model to relate drug exposure to prophylactic efficacy using standard statistical methods such as CART or non-linear regression. Summary statistics were also provided for the malaria incidence rate by cohort and treatment arm

SECONDARY OUTCOMES:
Number of subjects with adverse events, serious adverse events, and death | From screening to Day 43
  All information obtained on adverse events will be displayed by arm, treatment, and subject. The number and percentage of subjects with adverse events will be tabulated by body system and preferred term with a breakdown by cohort and treatment.
Pharmacokinetics of KAF156: Area under the plasma concentration-time curve from time zero to infinity (AUCinf) | Pre-dose, and Post-dose: 1 hour, 3 hours, 6 hours, 9 hours, 12 hours, 24 hours, 96 hours, 144 hours, 110 hours, 216 hours, 240 hours
  KAF156 plasma concentration data will be listed by arm, subject, and sampling time point.
  Descriptive summary statistics will be provided by arm and sampling time point. These values will be used to calculate AUCinf
Pharmacokinetics of KAF156: Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) | Pre-dose, and Post-dose: 1 hour, 3 hours, 6 hours, 9 hours, 12 hours, 24 hours, 96 hours, 144 hours, 110 hours, 216 hours, 240 hours
  KAF156 plasma concentration data will be listed by arm, subject, and sampling time point.
  Descriptive summary statistics will be provided by arm and sampling time point. These values will be used to calculate AUClast
Pharmacokinetics of KAF156: Area under teh plasma concentration-time curve from time zero to time 24 h (AUC0-24) | Pre-dose, and Post-dose: 1 hour, 3 hours, 6 hours, 9 hours, 12 hours, 24 hours, 96 hours, 144 hours, 110 hours, 216 hours, 240 hours
  KAF156 plasma concentration data will be listed by arm, subject, and sampling time point.
  Descriptive summary statistics will be provided by arm and sampling time point. These values will be used to calculate AUC0-24
Pharmacokinetics of KAF156: Terminal elimination half life (T1/2) | Pre-dose, and Post-dose: 1 hour, 3 hours, 6 hours, 9 hours, 12 hours, 24 hours, 96 hours, 144 hours, 110 hours, 216 hours, 240 hours
  KAF156 plasma concentration data will be listed by arm, subject, and sampling time point.
  Descriptive summary statistics will be provided by arm and sampling time point. These values will be used to calculate T1/2.
Pharmacokinetics of KAF156: Apparent systemic clearance from plasma following oral administration (CL/F) | Pre-dose, and Post-dose: 1 hour, 3 hours, 6 hours, 9 hours, 12 hours, 24 hours, 96 hours, 144 hours, 110 hours, 216 hours, 240 hours
  KAF156 plasma concentration data will be listed by arm, subject, and sampling time point.
  Descriptive summary statistics will be provided by arm and sampling time point. These values will be used to calculate CL/F
Pharmacokinetics of KAF156: Apparent volume of distribution during the terminal phase following oral administration (Vz/F) | Pre-dose, and Post-dose: 1 hour, 3 hours, 6 hours, 9 hours, 12 hours, 24 hours, 96 hours, 144 hours, 110 hours, 216 hours, 240 hours
  KAF156 plasma concentration data will be listed by arm, subject, and sampling time point.
  Descriptive summary statistics will be provided by arm and sampling time point. These values will be used to calculate Vz/F
Pharmacokinetics of KAF156: Observed maximum plasma concentration (Cmax) | Pre-dose, and Post-dose: 1 hour, 3 hours, 6 hours, 9 hours, 12 hours, 24 hours, 96 hours, 144 hours, 110 hours, 216 hours, 240 hours
  KAF156 plasma concentration data will be listed by arm, subject, and sampling time point.
  Descriptive summary statistics will be provided by arm and sampling time point. These values will be used to calculate Cmax
Pharmacokinetics of KAF156: Time to reach the maximum concentration (Tmax) | Pre-dose, and Post-dose: 1 hour, 3 hours, 6 hours, 9 hours, 12 hours, 24 hours, 96 hours, 144 hours, 110 hours, 216 hours, 240 hours
  KAF156 plasma concentration data will be listed by arm, subject, and sampling time point.
  Descriptive summary statistics will be provided by arm and sampling time point. These values will be used to calculate Tmax
Parasite growth Kinetics by qRT-PCR | Pre-dose, days 7-23, Day 29, Day 43
  Parasitemia levels as measured by qRT-PCR will be summarized and displayed graphically over time.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Seattle, Washington, United States

REFERENCES:
- [Derived] Kublin JG, Murphy SC, Maenza J, Seilie AM, Jain JP, Berger D, Spera D, Zhao R, Soon RL, Czartoski JL, Potochnic MA, Duke E, Chang M, Vaughan A, Kappe SHI, Leong FJ, Pertel P, Prince WT; KAF156 Study Team. Safety, Pharmacokinetics, and Causal Prophylactic Efficacy of KAF156 in a Plasmodium falciparum Human Infection Study. Clin Infect Dis. 2021 Oct 5;73(7):e2407-e2414. doi: 10.1093/cid/ciaa952. PMID 32644127